CLINICAL TRIAL: NCT00417846
Title: Age-related Macular Degeneration: Detection of Onset of New Choroidal Neovascularization (AMD DOC Study)
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Emily W. Gower, PhD, Johns Hopkins University
Other Study IDs: NA_00006147
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Maculopathy, Age-Related; Choroidal Neovascularization
Keywords: Age-Related Macular Degeneration; Optical Coherence Tomography, OCT; Preferential Hyperacuity Perimeter, PHP; Amsler Grid
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the sensitivity of the optical coherence tomography (OCT) test in detecting neovascular AMD in eyes at high risk for CNV development. In order to test this hypothesis, we are conducting a multi-center clinical study at four participating clinical centers. A total of 227 participants will be enrolled. Participants will be followed-up for a period of two years, or until CNV develops in the study eye for which treatment is recommended, to determine the occurrence of CNV. The fundamental design principles of the study are simplicity and parsimony.

DETAILED DESCRIPTION:
Primary Objective:

The purpose of this study is to determine the sensitivity of the OCT in detecting conversion to neovascular AMD by two years in eyes at high risk for CNV, with FA serving as the gold standard.

Secondary Objectives:

* To determine the specificity, positive predictive value, and negative predictive value of the OCT in detecting conversion to neovascular AMD by two years in eyes at high risk for CNV, with FA serving as the gold standard.
* To compare the sensitivity, specificity, positive predictive value, and negative predictive value of the OCT to the PHP or the supervised Amsler Grid in subjects who had either negative PHP and/or negative supervised Amsler grid at baseline for detection of neovascular AMD by two years in eyes at high risk for CNV
* To describe features of false positives and false negatives with respect to baseline characteristics seen on PHP testing, supervised Amsler grid testing, and OCT imaging
* To describe the relationship between new visual symptoms experienced by participants prompting an interim evaluation where treatment for CNV was recommended and findings seen at the previous study visit (PHP testing, supervised Amsler grid testing, OCT imaging, other findings on exam, or fluorescein angiography) as well as findings from the baseline visit
* To determine the physician's detection of CNV development on return study visits including slit lamp biomicroscopy before viewing ancillary tests from that visit (supervised Amsler grid, PHP, OCT, fundus photographs, fluorescein angiogram)

All participants will be examined upon enrollment and then followed every three months after enrollment for two years or until conversion to CNV is positive and treatment is recommended. Specifically, follow-up visits will occur at 3, 6, 9, 12, 15, 18, 21, and 24 months from the date of the Initial Visit.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age 50 years or greater
* Best corrected visual acuity letter score = 65 or greater (approximate Snellen equivalent of 20/50 or better in the candidate study eye)
* Neovascular AMD in the fellow eye and no CNV in the candidate study eye (absence of CNV confirmed by FA which will be graded in a masked fashion by the AMD DOC Study Reading Center)
* Candidate study eye must have evidence of at least one large druse (≥ 125µm) and focal hyperpigmentation within 3600μm of the fovea and visible on color fundus photography, red-free photograph, or fluorescein angiography
* Participant must have media clear enough in the candidate study eye to permit fundus photography, fluorescein angiography, and optical coherence tomography and absence of any fluorescein allergies
* Results of the baseline PHP and supervised Amsler grid will not affect eligibility of the participant. Subjects can be eligible for further follow-up even if they have positive PHP and Amsler grid
* Eligible participants who have a positive PHP or supervised Amsler grid for that eye at the initial screening visit should have a second PHP or supervised Amsler grid screening visit within 2 weeks in order to repeat the PHP or Amsler test or the participant may repeat the PHP or Amsler grid that day before pupillary dilation. Participants with a 2nd positive PHP or supervised Amsler grid are still eligible for further follow-up
* All tests (supervised Amsler grid, PHP, OCT, FA) must be performed within 2 weeks of each other
* Participants with non-foveal geographic atrophy in the candidate study eye are still eligible for enrollment in the study

Exclusion Criteria:

* Known allergy to fluorescein angiography or allergic reaction during screening
* Advanced AMD with CNV in both eyes confirmed on FA graded by the AMD DOC Study Reading Center
* Foveal geographic atrophy in the study eye
* Positive OCT test for the candidate study eye, as read by the AMD DOC Study Reading Center, for subretinal fluid, intraretinal edema, or retinal thickening that falls within the top 1% of the normative data base for the Stratus OCT
* Significant media opacity that precludes reasonable quality retinal imaging including color fundus photographs, fluorescein angiography, or OCT in the candidate study eye to assess the presence of CNV
* Evidence of macular disease (e.g., pattern dystrophy, diabetic macular edema, vitreomacular traction) other than AMD in the study eye
* Previous surgical or laser treatment to the macula of the study eye
* Diabetic retinopathy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have neovascular AMD in the fellow eye and non-neovascular AMD in the candidate study eye to be eligible for this study. Additional inclusion and exclusion criteria are listed below.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana V. Do, M.D., Study Chair — Johns Hopkins Medical Institutes; Neil M. Bressler, M.D., Study Director — Johns Hopkins Medical Institutes
Locations (4):
- United States (4):
  - Retina Vitreous Associates, Beverly Hills, California
  - The Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Associates of Cleveland, Beachwood, Ohio